CLINICAL TRIAL: NCT00964938
Title: Multisite Pacing With a Quadripolar Left Heart Lead in Cardiovascular Resynchronization Therapy (CRT) Patients
Brief Title: Multisite Pacing With a Quadripolar Lead
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MSLV
Record Dates: First submitted 2009-05-25; First posted 2009-08-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Hemodynamic response; Cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Quadripolar LV lead (pacing configurations) — Quadripolar LV lead will be used to deliver a combination of pacing configurations

SUMMARY:
The purpose of this study is to evaluate the effects of multisite left ventricular (LV) biventricular (BiV) pacing on LV hemodynamics in CRT patients. It is hypothesized that the effect of simultaneous BiV pacing utilizing multisite LV pacing on LV hemodynamics will be superior to conventional BiV pacing.

ELIGIBILITY:
Inclusion Criteria:

* Have a scheduled CRT implantation at the participating clinical study site
* Have NYHA functional class III or IV, ejection fraction less than or equal to 35%, and QRS duration greater than 120ms
* Be undergoing a new St. Jude Medical CRT-D device system (including LV lead) implantation
* Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed perioperative evaluations

Exclusion Criteria:

* Have persistent or permanent atrial fibrillation
* Have an intrinsic heart rate of <50 beats per minute
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures
* Have had a recent CVA or TIA within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Have ischemic etiology and are unable to tolerate stress echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
dP/dt max | acute: during implant procedure; 1 day

CONTACTS AND LOCATIONS:
Overall Officials: B Thibault, Principal Investigator — Montreal Heart
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Thibault B, Dubuc M, Khairy P, Guerra PG, Macle L, Rivard L, Roy D, Talajic M, Karst E, Ryu K, Paiement P, Farazi TG. Acute haemodynamic comparison of multisite and biventricular pacing with a quadripolar left ventricular lead. Europace. 2013 Jul;15(7):984-91. doi: 10.1093/europace/eus435. Epub 2013 Feb 27. PMID 23447571